CLINICAL TRIAL: NCT00325338
Title: Follow-up Study to Evaluate the Sustained Clinical Efficacy of Ragweed MATA MPL (Allergy Therapeutics®) in Patients With Ragweed-induced Seasonal Allergic Rhinitis Upon Re-exposure to Ragweed Pollen in an Environmental Exposure Chamber (EEC) Model, Approximately One Year After Pre-seasonal Treatment in 2005
Brief Title: Follow-up Investigation of Efficacy of Ragweed MATAMPL,and Placebo in Patients With Ragweed-induced Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RagweedMATAMPL205; P2DP05007
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy; Ragweed; Environmental Exposure Chamber
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Ragweed MATAMPL

SUMMARY:
Ragweed MATAMPL has been developed to provide pre-seasonal specific immunotherapy for patients with hypersensitivity to ragweed pollen (hay fever). This novel formulation is designed to provide a vaccine that will be efficacious with only four escalating dose injections administered before the start of the pollen season. In this Follow-up Study the Efficacy will be assessed by exposing allergic subjects to Ragweed pollen in an environmental exposure chamber EEC. Patient symptomatic response to pollen and patient quality of life in the EEC will be determined. Patients who previously completed two EEC portions of study Ragweed MATAMPL 204 and who had been treated with either Ragweed MATA MPL or Placebo before the 2005 ragweed season will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed both EEC periods of study P2DP5001; have had received either placebo or the top dose if they had been treated with Ragweed MATA MPL; and have had no major changes in medical history or health status since completing the study.
* Patients must be willing and able to give written informed consent and provide this consent prior to initiation of any study procedures, including initiation of washout of any concomitant medications.
* Patients must be willing and able to attend all study visits.
* Patients must observe the drug washout times listed in Table 3.2.3 prior to Screening (Visit 1). The use of other concomitant medications will be permitted if they are not expected to interfere with the ability of the patient to participate in the study and provided that they have been on a stable regimen (i.e. the same dose and schedule of administration) for eight weeks prior to screening).
* Women of childbearing potential must be using one of the following acceptable birth control methods:

  1. Intrauterine device (IUD) in place for at least three months;
  2. Barrier method (condom or diaphragm) with spermicide;
  3. Stable hormonal contraceptive for at least three months prior to study and through study completion;
  4. Abstinence;
  5. Not-heterosexual lifestyle.
* Patients must be able to follow instructions

Exclusion Criteria:

* Symptomatic for allergic rhinitis or allergic conjunctivitis from allergy to grass or trees at Visit 1.
* Symptomatic for significant perennial rhinitis at Visit 1, as judged by the Investigator.
* Concurrent disease that might complicate or interfere with investigation or evaluation of the study medication such as:
* Chronic use of antihistamines and other concomitant medications (e.g. tricyclic antidepressants) that would affect assessment of the effectiveness of study drug.
* Any systemic disorder that could interfere with the evaluation of the study medication.
* Upper or lower respiratory tract infection requiring antibiotics with 14 days of Visit 2.
* Diagnosis of sinusitis within 30 days of Visit 2.
* Any ocular disorder (other than allergic conjunctivitis) including presumed infectious ocular disease (bacterial, fungal, viral, etc.), which could interfere with the evaluation of the study drug.
* Hypersensitivity to the study drug excipients.
* Patients with active or quiescent tuberculous infection of the respiratory tract, untreated local or systemic fungal infection or bacterial or systemic viral infections or parasitic or ocular herpes simplex.
* Patients who have experienced nasal ulcers, nasal surgery or nasal trauma within 90 days of enrollment into this study.
* Clinical history of anaphylaxis or idiopathic anaphylaxis.
* Patients with contraindications for allergy vaccines.
* Patients with a clinical history of immunodeficiency, including those who are on immunosuppressant therapy.
* Patients in whom tyrosine metabolism is disturbed, especially in the case of tyrosinemia and alkaptonuria.
* Patients with contraindication to adrenaline.
* Subjects who are taking β-blockers for any indication including eye drops.
* Current diagnosis of chickenpox or measles.
* Clinical history of drug or alcohol abuse, at the Investigator's discretion, that would interfere with the patient's participation in the study.
* Clinical history of severe or uncontrolled cardiovascular, hepatic, renal and/or other diseases/illness that could be expected to interfere with the study.
* Clinical history, or evidence, of nasolacrimal drainage system malfunction.
* Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol.
* Patient who have participated in any other investigational study within 30 days of Visit 1 or concomitant with this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-05; Study Completion 2006-07

PRIMARY OUTCOMES:
to assess whether the efficacy of RagweedMATAMPL is maintained approximately one year later during the first EEC period of 2006

SECONDARY OUTCOMES:
Determine whether the lack of efficacy observed for Ragweed MATA MPL in 2005 will manifest itself approximately one year later
Determine whether the immunoglobulin levels measured after treatment with Ragweed MATA MPL in 2005 have changed approximately one year later.
Determine whether the responses to the RQLQ-EEC measured after treatment with Ragweed MATA MPL in 2005 have changed approximately one year later.
Determine whether a second treatment in 2006 will modify the efficacy observed in 2005 and maintained approximately one year later in patients who had been treated with Ragweed MATA MPL.
Determine whether a second treatment in 2006 will modify the efficacy observed in 2005 and partially or completely lost approximately one year later in patients who had been treated with Ragweed MATA MPL
Determine whether a second treatment in 2006 will confer or improve the efficacy in patients who moderately responded or did not respond to Ragweed MATA MPL in 2005
Determine whether a second treatment in 2006 will modify the extent of the immunoglobulin response observed in 2005 in patients who had been treated with Ragweed MATA MPL
Determine whether a second treatment in 2006 will modify the responses to the RQLQ-EEC recorded before and after treatment in 2005

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International Inc.
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada